CLINICAL TRIAL: NCT03362112
Title: Lipoprotein-associated Phospholipase A2 in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ENDO20171130-1
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Results first posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2017-11

CONDITIONS: Type2 Diabetes
Keywords: lipoprotein-associated phospholipase A2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lipoprotein-associated phospholipase A2 (LP-PLA2) is a good marker of cardiovascular risk and inflammation. This study aims at the characteristic and clinical significance of LP-PLA2 test in patients with type 2 diabetes(T2D).

DETAILED DESCRIPTION:
The investigators recorded clinical factors, serum levels of glucose, HbA1c, lipids and LP-PLA2 in patients with T2D who visited in the Department of Endocrinology at the Nanjing First Hospital from January 2015 to August 2016. The relationship between levels of LP-PLA2 and diabetic complications are analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2D and the diagnostic criteria of T2D is according to the World Health Organization in 1999.

Exclusion Criteria:

1. Patients use systemic steroidal anti-inflammatory drugs.
2. Patients are pregnant.
3. Patients with an acute infection.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with type 2 diabetes who visited in the Department of Endocrinology at the Nanjing First Hospital from January 2015 to August 2016 were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 1713 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2017-06-01 (Actual)

REFERENCES:
- [Derived] Hu Y, Li TT, Zhou W, Lu TT, Li FF, Ding B, Liu BL, Xie XJ, Ma JH. Lipoprotein-associated phospholipase A2 is a risk factor for diabetic kidney disease. Diabetes Res Clin Pract. 2019 Apr;150:194-201. doi: 10.1016/j.diabres.2019.03.026. Epub 2019 Mar 20. PMID 30904742

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With T2DM: Patients with type 2 diabetes
Period: Overall Study
Arm/Group | Patients With T2DM
Started | 1713
Completed | 1622
Not Completed | 91

BASELINE CHARACTERISTICS:
Arm/Group | Patients With T2DM
Number analyzed (Participants) | 1713
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 658
  Male | 1055
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  China | 1713

OUTCOME MEASURES:

1. Primary Outcome: Lipoprotein-associated Phospholipase A2
Description: the plasma lipoprotein-associated phospholipase A2 level of patients
Time Frame: Day one
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Patients With T2DM
Number analyzed (Participants) | 1452
ng/ml | 238.4 (111.9)

2. Secondary Outcome: HbA1c
Description: the glycosylated hemoglobin level of patients
Time Frame: Day one
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Patients With T2DM
Number analyzed (Participants) | 1452
percentage of glycated hemoglobin | 9.1 (2.1)

3. Secondary Outcome: LDL-c
Description: low density lipoprotein cholesterol
Time Frame: Day one
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Patients With T2DM
Number analyzed (Participants) | 1452
mmol/L | 2.5 (0.8)

4. Secondary Outcome: Diabetic Complication
Description: the prevalence of atherosclerosis, diabetic Nephropathy, diabetic retinopathy and diabetic neuropathy
Time Frame: Day one
Reporting Status: Not Posted

5. Secondary Outcome: C Peptide
Description: fast and 120min postprandial C peptide
Time Frame: Day one
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Serious, and Other Adverse Events were not assessed.
Arm/Group | Patients With T2DM
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes